CLINICAL TRIAL: NCT06870773
Title: Impact of Helicobacter Pylori Infection on Prolactin Levels in Reproductive-Age Women in Upper Egypt
Brief Title: Impact of Helicobacter Pylori Infection on Prolactin Levels in Reproductive-Age Women to Determine Whether H. Pylori Infection is Associated with Elevated Prolactin Levels and Assess the Clinical Implications
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandra Maged Ezzat Rasmi, resident at the internal medicine department, Assiut University
Other Study IDs: Impact of Hpylori on prolactin
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Hyperprolactinaemia
Keywords: H.pylori; prolactin level; hyperprolactinemia
MeSH Terms: conditions — Hyperprolactinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- H. pylori-positive reproductive-age women: This group consists of women aged 18-45 years with confirmed H. pylori infection, as determined by stool antigen tests or breath tests and IgM serum. Participants are within reproductive age, not currently pregnant or breastfeeding, and have no known endocrine disorders or chronic illnesses that could affect prolactin levels. The study will measure their serum prolactin levels to investigate the potential association between H. pylori infection and hyperprolactinemia, as well as assess related reproductive health outcomes.

SUMMARY:
The research is a cross-sectional observational study conducted at Assiut University Hospital. It will involve 75 women aged 18-45 with confirmed H. pylori infection. The study will measure serum prolactin levels and H. pylori infection status through stool antigen tests. The primary outcome is comparing prolactin levels between H. pylori-positive and negative women. Secondary outcomes include analyzing correlations with clinical symptoms and demographic factors.

DETAILED DESCRIPTION:
Study Design and Setting Cross-sectional observational study

Conducted at Assiut University Hospital

Sample size: 75 women

Participants Inclusion criteria: Women aged 18-45, confirmed H. pylori infection, reproductive age

Exclusion criteria: Recent antibiotic or PPI use, endocrine disorders, chronic illnesses affecting prolactin

Data Collection Participant recruitment from outpatient clinics

Laboratory assessments:

Stool antigen test for H. pylori using ELISA method

Serum prolactin measurement via chemiluminescent immunoassay

Questionnaire for demographic information and medical history

Outcome Measures Primary: Serum prolactin levels in H. pylori-positive vs. negative women

Secondary: Correlation with clinical symptoms and demographic factors

Analysis The study will compare prolactin levels between H. pylori-positive and negative groups, analyze correlations with symptoms, and assess the influence of demographic factors on prolactin levels and H. pylori prevalence.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age Range: Women aged 18 to 45 years. 2. Diagnosis of H. pylori Infection: Participants must have a confirmed diagnosis of H. pylori infection through non-invasive methods such as stool antigen tests or breath tests and IgM serum.

3. Reproductive Age: Women must be within reproductive age and not currently pregnant or breastfeeding

Exclusion Criteria:

* 1. Recent Antibiotic Use: Individuals who have taken antibiotics within the last month will be excluded to avoid interference with H. pylori detection.

  2. Use of Proton Pump Inhibitors (PPIs): Patients using PPIs or other medications that affect gastric acid secretion within the last month will be excluded.

  3. Endocrine Disorders: Women with known endocrine disorders such as hyperprolactinemia from other causes will be excluded.

  4. Chronic Illnesses: Individuals with chronic illnesses that could affect prolactin levels (e.g., renal failure, liver disease) will also be excluded.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 45 years and confirmed diagnosis of H. pylori infection through non-invasive methods such as stool antigen tests or breath tests and IgM serum.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Prolactin Levels: | 1 month
  Prolactin Levels: The primary outcome measure will be the serum prolactin levels in women diagnosed with H. pylori infection compared to those without infection.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 8. Chittajallu RS, Doraiswamy S, Prakash K, Babu S. Helicobacter pylori infection and its association with hyperprolactinemia: a cross-sectional study. J Clin Diagn Res. 2020;14(3):OC01-OC04.